CLINICAL TRIAL: NCT00470925
Title: Assessment of the Effect of Sertaline on the Specific Binding of 123-I MZINT in Healthy Subjects
Acronym: mZINT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: mZINT_003
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: Neurological; Dopamine
MeSH Terms: conditions — Depression; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access [123I]MZINT and SPECT Imaging (Experimental)
  Interventions: Drug: 123-I MZINT injection and SPECT imaging

INTERVENTIONS:
Drug: 123-I MZINT injection and SPECT imaging — SPECT imaging uses the single photon emissions from radioactive compounds that are (most commonly) injected into a patient and are metabolized by specific organs or body systems. SPECT imaging is performed by using a gamma camera to acquire multiple 2-D images (also called projections), from multiple angles. A computer is then used to apply a tomographic reconstruction algorithm to the multiple projections, yielding a 3-D dataset. This dataset may then be manipulated to show thin slices along any chosen axis of the body, similar to those obtained from other tomographic techniques, such as MRI, CT, and PET. The resulting SPECT images reflect body/organ function as opposed to specific anatomy of other imaging modalities such as CT or MRI

SUMMARY:
The overall purpose of this project is to evaluate the effect of sertraline administration on the binding of 123-I mZINT in 10 healthy subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT.

DETAILED DESCRIPTION:
Serotonin (5-HT) is a monoamine neurotransmitter found in the peripheral and central nervous system. It is responsible for regulating a wide variety of physiological processes and higher CNS functions. 5-HT neurons project diffusely throughout the brain, innervating the cerebral cortex, hippocampus, thalamus, midbrain, brainstem and cerebellum, and play a prominent role in regulating physiological and behavioral responses such as arousal, thermoregulation, anxiety, and affect.

All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, and a baseline physical and neurological evaluation. healthy subjects will undergo a baseline 123-I MZINT injection and SPECT imaging described below. At baseline, healthy subjects will be started on either no treatment (n=4), or one of three different doses of sertraline (25 mg/day n=2, 50 mg/day n=2 or 150 mg/day n=2), which will be administered over a 14 day period. Fourteen days following imaging session 1, all subjects (treated with sertraline and untreated) will undergo a second 123-I MZINT and SPECT imaging study. Data from the baseline and follow-up SPECT images will be compared to evaluate for any effect of sertraline on regional brain uptake of 123-I MZINT. The subjects that are randomized to no treatment will serve as controls and provide preliminary test-retest reproducibility data on the imaging outcome measure.

The goal of this proposal is to evaluate the effect of sertraline administration on the specific [123-I] mZINT. In vitro and in vivo data from early human studies and baboon studies strongly support further evaluation of [123I] mZINT in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 18-70.
* Written informed consent is obtained.
* The participant has no clinically significant clinical laboratory value and/or clinically significant unstable medical, neurological or psychiatric illness.
* For females, non-child bearing potential or negative urine pregnancy test on day of [123I] mZINT injection.
* Willingness to comply with the study protocol

Exclusion Criteria:

* The subject has a clinically significant clinical laboratory values abnormality, and/or medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Use of all prescription drugs or non-prescriptions drugs that may effect serotonin such as antidepressants including sertraline, fluoxetine, fluvoxamine, venlafaxine within 60 days of baseline imaging study.
* The participant has a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM IV) {American Psychiatric Association, 1994 #2} within the past 2 years.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Does administration of sertraline have an effect on the specific binding of 123-mZINT in healthy subjects evaluated with serial, dynamic SPECT imaging at baseline and after 14 days of sertraline treatment? | 14 DAYS

SECONDARY OUTCOMES:
Is there a dose effect of sertraline on 123I MZINT binding? Do higher doses of sertraline have a more profound effect on the specific binding of 123I MZINT than lower doses of sertraline? | 14 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Danna L. Jennings, MD, Principal Investigator — unafilliated
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Brooks DJ, Piccini P. Imaging in Parkinson's disease: the role of monoamines in behavior. Biol Psychiatry. 2006 May 15;59(10):908-18. doi: 10.1016/j.biopsych.2005.12.017. Epub 2006 Apr 11. PMID 16581032
- See also: IND web page — http://www.indd.org
- See also: MNI web page — http://www.mnimaging.com